CLINICAL TRIAL: NCT04821141
Title: Randomized IIB Study of the Effect of Bazedoxifene Plus Conjugated Estrogens on Breast Imaging and Tissue Biomarkers in Peri or Post-Menopausal Women at Increased Risk for Development of Breast Cancer
Brief Title: Phase IIB Trial of Bazedoxifene Plus Conjugated Estrogens
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Carol Fabian, MD, Professor, University of Kansas Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00146320; R01CA249437 (NIH)
Record Dates: First submitted 2021-03-18; First posted 2021-03-29 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Risk Reduction; Breast Cancer
Keywords: breast cancer, menopausal symptoms, hot flashes
MeSH Terms: conditions — Risk Reduction Behavior; Breast Neoplasms; Hot Flashes | interventions — bazedoxifene; Estrogens, Conjugated (USP)

STUDY DESIGN:
Intervention Model Description: Randomization to immediate 6 months of BZA+CE versus wait list for 6 months followed by option to receive 6 months of BZA+CE.
Masking Description: Only designated biostatistician is aware of randomization assignment until after a subject is enrolled and assigned, Then assignment is unblinded and agents are open-label.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Bazedoxifene plus conjugated estrogens immediately (Experimental): BZA (20 mg) plus CE (0.45 mg) taken together once daily for 6 months, commencing immediately.
  Interventions: Drug: Bazedoxifene and Conjugated Estrogens
- Bazedoxifene plus conjugated estrogens wait list (Other): No intervention for initial 6 months (wait list), then BZA (20 mg) plus CE (0.45 mg) taken together once daily for 6 months, commencing 6 months after enrollment. Optional on the part of subject.
  Interventions: Drug: Bazedoxifene and Conjugated Estrogens

INTERVENTIONS:
Drug: Bazedoxifene and Conjugated Estrogens — BZA (20 mg) plus CE (0.45 mg) taken together once daily
  Other Names: BZA+CE

SUMMARY:
Women at risk for development of breast cancer and experiencing vasomotor menopausal symptoms (hot flashes) will be randomized to bazedoxifene (BZA) plus conjugated estrogens (CE) for 6 months versus a wait list control. Two risk factors for development of breast cancer will be studied pre-study and after 6 months: fibroglandular volume (FGV) on mammogram as assessed by Volpara software and proliferation by Ki-67 immunocytochemistry in benign breast tissue acquired by random periareolar fine needle aspiration (RPFNA). Change in biomarkers will be compared between groups.

DETAILED DESCRIPTION:
Phase IIB trial of 6 months of BZA 20 mg +CE 0.45 mg (subsequently designated as BZA+CE) vs a waitlist control. Trial is informed by prior results of a single arm trial that used Duavee® (combination of BZA+CE that is FDA-approved for relief of hot flashes). Since Duavee® is currently not available commercially, the two separate components are used instead. Breast imaging, benign breast tissue by RPFNA, and blood for biomarkers will be obtained at baseline and at 6 months using similar assessment techniques. The primary endpoint is the difference between the BZA+CE and control groups for absolute change from baseline to 6 months in the risk biomarker fibroglandular volume (FGV). Volpara® fully automated assessments overcome the interpretive variance inherent in subjective assessments. Additional endpoints include changes in benign breast epithelial immunolabeling for Ki-67, estrogen receptor alpha (ERα), progesterone receptor (PR), and anterior gradient-2 protein (AGR2); and systemic levels of bioavailable hormones, IGF-1, IGFBP3, and measures of insulin sensitivity. The modifying effects of baseline BMI, visceral adipose, and plasma BZA concentrations on markers will be studied.

ELIGIBILITY:
Inclusion Criteria for Baseline Mammogram and RPFNA Women ages 45 - 60 or ages 61-64 if their last mammogram was described as heterogeneously or extremely dense.

Current vasomotor symptoms (hot-flashes, night sweats or both). These do not need to be frequent or severe but should occur at least once a week. Women who feel that they would likely need a supplement or be at high risk of withdrawal if they were randomized to waitlist because of vasomotor symptoms are not good candidates for this trial.

Women must be in one of the four menopausal status categories, as defined below.

* Age 45-64 with an intact uterus and no periods in past 12 months. Amenorrhea is not thought to be due to endometrial ablation, Mirena IUD or other menses suppressing contraceptives. Category 1: Clinically Postmenopausal
* Age 45-64 with an intact uterus and no periods in past 2 months immediately preceding eligibility testing; but has not been amenorrheic for 12 months. Amenorrhea not thought to be due to endometrial ablation, Mirena IUD or other menses suppressing contraceptives. Category 2: Late menopause transition.
* Age 50-64 and prior hysterectomy, prior endometrial ablation with subsequent lack of periods, or menses suppression due to Mirena IUD or other types of contraceptives. Category 3: Menopause transition by symptoms; uterus not intact or menses suppression; age ≥50.
* Age 45-49 and prior hysterectomy, prior endometrial ablation with subsequent lack of periods, or menses suppression due to Mirena IUD or other types of contraceptives. Category 4: Menopause transition by symptoms uterus not intact or menses suppression; age 45-49.

Must have at least one ovary.

BMI: ≤ 38 kg/m2

At least one breast without prior therapeutic radiation that can be assessed by Volpara® software.

Chemistry profile showing reasonably normal renal and hepatic function: creatinine <2.0 mg/dL, bilirubin < 2.5 mg/dL, and albumin > 3.4 g/dL within the past 12 months.

Risk Factors/Level. Moderate risk of developing breast cancer based on having at least one of following:

* First or second degree relative with breast cancer age 60 or younger;
* A prior breast biopsy showing proliferative breast disease, including hyperplasia, atypical hyperplasia, or lobular carcinoma in situ
* 2 or more prior biopsies regardless of benign histology
* Prior ER-PR- or low risk ER+ DCIS at minimum treated with surgical removal of lesion with or without radiation therapy.
* Surgical removal of DCIS is defined as no DCIS cells within 2 mm of the margin or if DCIS cells were present at the margin, a subsequent resection shows no DCIS cells and there were no residual calcifications on the mammogram.
* Low risk ER+ and/or PR+ DCIS is defined as that which is ≤2 cm in diameter, non-high grade and occurring in women who are 50 or older.
* Women with known gene mutations associated with an increased risk for breast cancer such as ATM, CDH1, CHEK2, NBN, NF1, PALB2, PTEN, STK11, P53, PTEN (Note: BRCA1/2 are excluded as women 45 and over should have undergone risk-reducing bilateral salpingo-oophorectomy).
* 10-year relative risk of ≥2X that for the average population for age group as calculated by IBIS Breast Cancer Risk Evaluation Tool version 8 (Tyrer-Cuzick) (http://www.ems-trials.org/riskevaluator/); or 10 year risk based on the Breast Cancer Surveillance Consortium tool Version 2 (https://tools.bcsc-scc.org/BC5yearRisk/calculator.htm)

Vaginal Hormones: Low dose vaginal hormones, such as Estring(®, Vagifem®, Imvexy®, or 0.5 gram or less of conjugated estrogen vaginal cream twice weekly or less often, for vaginal dryness and dyspareunia may be continued at the same dose.

Systemic Hormones: If previously on oral contraceptives or systemic hormone replacement such as pills, transdermal patches, oral troches, or injections, must be off for 8 weeks or more prior to baseline mammogram and RPFNA.

Exclusion Criteria for Screening

Conditions:

* Have a predisposition to or prior history of thromboembolism, deep venous thrombosis, pulmonary embolism, stroke, or myocardial infarction. Note that individuals with a prior septic embolus only with no evidence of a clotting disorder are not excluded if cleared by their cardiologist or internist.
* Prior bilateral oophorectomy
* BRCA1/2 deleterious mutation
* LCIS specifically designated as pleomorphic in the pathology report
* Prior high-risk ER+ and/or PR+ DCIS, defined as high grade, > 2 cm in diameter or diagnosed at age < 50.
* Prior DCIS with cancer cells at inked margin where there was not an additional resection.
* Prior invasive breast cancer
* Prior invasive uterine or ovarian cancer
* Current renal or liver disease or clinically significant abnormalities of liver and renal function tests.
* Known hypoparathyroidism or recent history of triglycerides > 300 mg/dl.
* Women are sufficiently distressed by their vasomotor symptoms, such that they do not believe they would be able to remain on study for 6 months without additional medications if their hot flashes were not relieved.
* Any other condition or intercurrent illness that in the opinion of the investigator makes the woman a poor candidate for RPFNA or treatment with BZA+CE.

Medications

* Current anticoagulant use (must have discontinued for 3 weeks prior to FNA)
* Taking oral or transdermal systemic hormones within two months (eight weeks) prior to baseline blood, imaging studies or RPFNA. (Note that continued use of vaginal low dose hormonal preparations for dyspareunia is allowed if the woman had been on for at least 2 weeks prior to baseline testing)
* Taken tamoxifen, raloxifene, or an aromatase inhibitor within 6 months of baseline blood imaging or RPFNA

Inclusion Criteria for Randomization Study mammograms

* 3D mammograms must be performed within 3 months of RPFNA. Women whose breast size require mosaic views will not be eligible.
* Clinical mammogram Interpretation: Mammograms read out as Class 0 or IV must be resolved with additional procedures prior to randomization or entry on intervention phase. Women having a recent benign biopsy subsequent to a BIRADS IV mammogram with continuing BIRADs IV on baseline mammogram for Volpara assessment may be entered if other clinical assessments (i.e., MRI) is judged as not worrisome for cancer and/or re-biopsy or re-excision is not being considered by the patient's clinical team.
* Raw data DICOM files must be available for generation of Volpara Score Card. Study consent must be signed prior to sending the DICOM files to the researcher server as these files will contain patient identifiers.
* A Volpara score card must be generated for at least 1 breast and the FGV must meet minimal requirements for BMI.
* If BMI < 25 kg/m2, then FGV must average at least 20 cm3 per breast (i.e., ≥20 cm3 if only one breast evaluable and ≥40 cm3 total if both breasts evaluable).
* If BMI is 25-38 kg/m2 then FGV must be at least 30 cm3 per breast (i.e., ≥30 cm3 if only one breast evaluable and ≥60 cm3 total if both breasts evaluable).
* The Volpara® "Score Card" must be sent to KUMC prior to randomization.

RPFNA must be performed and specimen received at KUMC in good condition. RPFNA specimen must have ductal/lobular epithelial cells on Thinprep® slides; but there is no requirement for a specific cell number, value for Ki-67, or cytomorphology.

Blood must be drawn prior to randomization and sent to KUMC.

Complete Menopause specific quality of life questionnaire, information for hot flash score.

Willing to comply with study procedures.

Participants at KUMC: Dual energy x-ray absorptiometry (iDXA)

Pregnancy test for women <age 55 with intact uterus

Exclusion Criteria for Randomization Intercurrent illness which makes potential participant unsuitable for study; Starting hormone replacement therapy (prescription pills, injections, patches) between mammogram/RPFNA and enrollment on study.

Ages: 45 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-12-14 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in FGV | baseline to 6 months
  Change in fibroglandular volume assessed on 3-D digital mammogram by Volpara software.

SECONDARY OUTCOMES:
Change in proliferation | baseline to 6 months
  change in percent of breast epithelial cells staining positive for Ki-67 by immunocytochemistry

OTHER OUTCOMES:
Change in blood hormones | baseline to 6 months
  Exploratory analysis of change in levels of hormones (estradiol, progesterone, testosterone, sex hormone binding globulin, etc.) assessed by ELISA or RIA methods at baseline and at 6 months.
change in gene expression | baselne to 6 months
  Exploratory analysis of changes and patterns of change in levels of mRNA assessed by qRT-PCR

CONTACTS AND LOCATIONS:
Overall Officials: Carol J Fabian, MD, Principal Investigator — University of Kansas Medical Center
Locations (6):
- United States (6):
  - City of Hope Medical Center, Duarte, California
  - University of California San Francisco, San Francisco, California
  - Northwestern Medical Center, Chicago, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fabian CJ, Nye L, Powers KR, Nydegger JL, Kreutzjans AL, Phillips TA, Metheny T, Winblad O, Zalles CM, Hagan CR, Goodman ML, Gajewski BJ, Koestler DC, Chalise P, Kimler BF. Effect of Bazedoxifene and Conjugated Estrogen (Duavee) on Breast Cancer Risk Biomarkers in High-Risk Women: A Pilot Study. Cancer Prev Res (Phila). 2019 Oct;12(10):711-720. doi: 10.1158/1940-6207.CAPR-19-0315. Epub 2019 Aug 16. PMID 31420361
- [Background] Carroll TJ, Abernethy PJ, Logan PA, Barber M, McEniery MT. Resistance training frequency: strength and myosin heavy chain responses to two and three bouts per week. Eur J Appl Physiol Occup Physiol. 1998 Aug;78(3):270-5. doi: 10.1007/s004210050419. PMID 9721008